CLINICAL TRIAL: NCT06573775
Title: Evaluation of Pain Quality in Young Swimmers Suffering From Myofascial Pain Syndrome Using Lidocaine Phonophoresis: A Randomized Controlled Trial
Brief Title: Evaluation of Pain Quality in Young Swimmers Suffering From Myofascial Pain Syndrome Using Lidocaine Phonophoresis
Acronym: MPS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New Ismailia National University (Other)
Responsible Party: Principal Investigator, Mohamed Abdel Moeim Abo EL Ros, Lecturer of Physical Therapy for Pediatrics and its Surgeries, New Ismailia National University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/001708
Record Dates: First submitted 2024-08-19; First posted 2024-08-27 (Actual); Last update posted 2024-08-27 (Actual); Status verified 2024-08

CONDITIONS: Neck Pain
Keywords: Myofascial; phonophoresis; pain
MeSH Terms: conditions — Neck Pain; Pain | interventions — Myofascial Release Therapy

STUDY DESIGN:
Intervention Model Description: randomized controlled trial
Who Masked: Participant
Masking Description: sealed envelopes
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control group A (Active Comparator): the control group received the traditional physical therapy for treating myofascial trigger points in the form of a myofascial trigger point release, stretching and strengthening of the trapezius muscle
  Interventions: Other: myofascial release
- study group B (Experimental): received pulsed ultrasound in addition to traditional physical therapy for treating myofascial trigger points in the form of a myofascial trigger point release, range of motion exercises, stretching and strengthening of the trapezius muscle
  Interventions: Device: pulsed ultrasound; Other: myofascial release
- study group C (Experimental): received lidocaine hydrochloride gel 5%phonophoresis in addition to traditional physical therapy for treating myofascial trigger points in the form of a myofascial trigger point release,range of motion exercises stretching and strengthening of the trapezius muscle
  Interventions: Other: myofascial release; Device: lidocaine phonophoresis

INTERVENTIONS:
Device: pulsed ultrasound — treatment of myofacial trigger points with therapeutic ultrasound
  Arms: study group B
Other: myofascial release — manual massage and range of motion exercises
  Other Names: myofascial trigger point realease
Device: lidocaine phonophoresis — transdermal tranmission of lidocaine molecules via ultrasound
  Arms: study group C

SUMMARY:
To evaluate pain quality by pain quality assessment scale (PQAS) using lidocaine phonophoresis on myofascial pain syndrome (MPS) in athletic children.

DETAILED DESCRIPTION:
Forty five males athletic swimmer children (10 to 14 years old) with MPS in the upper trapezius muscle were evaluated before and after treatment. They were randomly divided into three groups, n=15 children each. A (control), B and C (study groups). The three groups received spatial designed physical therapy program. The two study groups received pulsed ultrasound and lidocaine phonophoresis repectively. The duration of treatment was 40 minutes, three times / weeks for three successive months.

ELIGIBILITY:
Inclusion Criteria:

* Age range from 10 to 14 years.
* All children have regional neck pain complaint.
* Tenderness in cervical trigger points in the midpoint of the upper border of trapezius muscle, from grade II to grade IV according to tenderness grading scheme (Hubbard and Berkoff, 1993) (Appendix I )
* The diagnosis of an active MTrP in the upper trapezius according to (Ardiçet al . , 2002 and Bruno, 2005):
* Patients suffered from active MTrPs in the upper trapezius.
* Tender spots in one or more palpable taut bands.
* A typical pattern of referred pain distributed in the ipsilateral, posterolateral cervical paraspinal area, mastoid process or temporal area
* Palpable or visible local twitch response on snapping palpation at the most sensitive spot in the taut band.
* Restricted range of motion in lateral bending of the cervical spine to the opposite side.
* Palpation of a trigger point elicits a stereotypic zone of referred pain specific to that muscle.
* Identification of a palpable taut band, as well as a palpable, and exquisitely tender spot along the length of that taut band.
* All children allowed to practice their regular sport activities.

Exclusion Criteria:

* Neurological disorders.
* Dermatological disorders.
* Acute trauma prior to the study.
* Fibromyalgia, systemic disease and drug allergy history were excluded from the study.
* Having myofascial trigger points injection.
* Chronic pain in both sides of the body.
* History of findings of cervical injury whether orthopedic or soft tissue injury

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — adolescents
Enrollment: 45 (Actual)
Dates: Start 2023-06-05 (Actual); Primary Completion 2024-05-10 (Actual); Study Completion 2024-07-29 (Actual)

PRIMARY OUTCOMES:
pain quality | 6 weeks
  pain quality assessment scale with zero indication of better outcome and twenty means the worst outcome

SECONDARY OUTCOMES:
serum cortisol level | 6 weeks
  measurement of serum cortisol level

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed AM El Meligy, MD, Study Chair — Suez Canal University
Locations (1):
- College of Medicine, Ismailia, Egypt

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form: statistical plan with brief description (2024-08-01): https://cdn.clinicaltrials.gov/large-docs/75/NCT06573775/Prot_SAP_ICF_000.pdf
  • Informed Consent Form: consent form with brief description (2024-08-01): https://cdn.clinicaltrials.gov/large-docs/75/NCT06573775/ICF_001.pdf